CLINICAL TRIAL: NCT02415634
Title: Investigation of Physiotherapy Led ICU Discharge Facilitation Using the REhabilitation After Critical Illness Assisted Discharge Pack (RECAP) Model; a Pilot Randomized Controlled Trial.
Brief Title: REhabilitation After Critical Illness Assisted Discharge Pack (RECAP)
Acronym: RECAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maire Gilmartin (Other)
Collaborators: University of Ulster (Other); St Vincent's University Hospital, Ireland (Other)
Responsible Party: Sponsor-Investigator, Maire Gilmartin, Senior Physiotherapist Critical Care, St Vincent's University Hospital, Ireland
Organization: St Vincent's University Hospital, Ireland (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GilmartinSept2014
Record Dates: First submitted 2015-04-06; First posted 2015-04-14 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-04

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention Participants in the experimental group will receive usual care plus the RECAP with ICU therapist follow up after ICU discharge. This will be provided for a period of 3 weeks after intensive care unit discharge.
  Interventions: Other: RECAP
- Control (Active Comparator): Control Patients (Controls) will not receive formal (study-related) rehabilitation interventions and will only receive usual care.
  Interventions: Other: Control

INTERVENTIONS:
Other: RECAP — Patients will receive an information pack at ICU discharge called the RECAP. This pack will include
  * Part 1: A critical care discharge summary (UCCDIP) (Bench and Day, 2012)
  * Part 2: A rehabilitation goal setting care plan
  * Part 3: A patient communication forum
  * Part 4: Useful supports and contact information
  * Part 5: Tailored exercise programme
  The patient will have a consultation with the ICU physiotherapist before ICU discharge once weekly thereafter for 3 weeks . The focus of the session will be to discuss goal attainment and associated challenges.
  The ICU therapist will meet once weekly with the patient's primary physiotherapist to provide clinical support if necessary, in determining the patient's needs post critical care.
  Arms: Intervention
Other: Control — Participants allocated to the control group will receive standard physiotherapy intervention post ICU discharge
  Arms: Control

SUMMARY:
The complexity of critical illness can result in both physical and psychological consequences for survivors, which can extend past the intensive unit care stay and after hospital discharge. A need for information and empowerment in the recovery process are highlighted for developing treatment strategies. It is suggested that there is a relationship between physical problems and psychological symptoms, but this has not been researched. This pilot study aims to test the effectiveness of a physiotherapy directed Rehabilitation after Critical illness Assisted discharge Pack (RECAP) on the physical and psychological function of patients recovering from critical illness in the first three weeks post discharge from ICU to the general ward area. The study will rely on a randomized controlled clinical trial design, with patients assigned to either a "usual care" control group vs. the treatment group. It is expected that engaging patients in their rehabilitation plan will focus physiotherapy treatment and improve physical recovery. It is hypothesized that the RECAP will reassure, support and empower patients to directly affect their psychological recovery in the first three weeks after critical illness.

DETAILED DESCRIPTION:
The process of recovering from critical illness is complex. The physical and psychological consequences of surviving critical illness can extend past the intensive unit care stay and after hospital discharge. For a critically ill patient, their first transition is being discharged from intensive care to a general ward and is one of the most stressful transitions they experience. They are required to adjust both physically and psychologically as they begin an uncertain journey to recovery. Research on the patient experience has identified vulnerability, hopelessness, fear of the unknown and anxiety as key features of this transition. A need for information and empowerment in the recovery process are highlighted for developing treatment strategies. It is suggested that there is a relationship between physical problems and psychological symptoms but this has not been researched. There is also limited evidence to guide clinicians in treatment strategy choice for these patients. This pilot study aims to test the effectiveness of a physiotherapy directed Rehabilitation after Critical illness Assisted discharge Pack (RECAP) on the physical and psychological function of patients recovering from critical illness in the first three weeks post discharge from the ICU to the general ward area. The study will rely on a randomized controlled clinical trial design, with patients assigned to either a "usual care" control group vs. the treatment group. Individuals in the treatment group will receive "usual care" plus a RECAP pack at ICU discharge with once weekly follow up with an ICU physiotherapist. The intervention group will receive the RECAP plus standard physiotherapy for the first three weeks after intensive care stay and the control group will receive standard physiotherapy alone. Outcome measures used will be the Functional Independence Measure (FIM) and State Anxiety Inventory (SAI). Secondary Outcome measures will include the Chelsea Critical Care Physical Assessment Tool (CPAx) and a 5 question patient satisfaction questionnaire. Outcome measures will be taken at ICU discharge, at one week post ICU discharge and at three weeks after ICU discharge to determine physical and psychological recovery, along with evaluating overall study feasibility. It is expected that engaging patients in their rehabilitation plan will focus physiotherapy treatment and improve physical recovery. It is hypothesized that the RECAP will reassure, support and empower patients to directly affect their psychological recovery in the first three weeks after critical illness.

The User Centred Critical Care Discharge Information Pack (UCCDIP) and instructions, designed by Bench and Day (2012), will be used as a component of the RECAP. These are being used with the authors permission.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to ICU >4 days
* Indication for physiotherapy referral in ICU
* Indication for follow up physiotherapy on discharge from the ICU
* Age>18 years
* RASS score 0 at time of consent

Exclusion Criteria:

* ICU length of stay >14 days
* Patients with a multi-disciplinary team based work-up in advance of a planned ICU admission (e.g. Liver transplant)
* Pregnant mothers
* Palliation
* Expected discharge to another hospital
* Unable to understand English
* Patients who have direct access to condition specific MDT follow up (e.g. Stroke, Neurology)
* Psychiatric Disease
* Unstable Cardiac Disease
* Where physiotherapy treatment is limited or maximal functional capacity is capped for duration of study (e.g. Non Weight Bearing status due to orthopaedic limitation x 12 weeks.
* Patients who are unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Functional Independence Measure (FIM) | Assessed at week three to detect change from baseline FIM score as a result of intervention
  A measure of physical and cognitive function
Change from baseline State Anxiety inventory (SAI), a subscale of State-Trait Anxiety Inventory | Assessed at week one to detect change from baseline in SAI score as a result of intervention
  A measure of state anxiety
Change from baseline State Anxiety inventory (SAI), a subscale of State-Trait Anxiety Inventory | Assessed at week three to detect change from baseline in SAI score as a result of intervention
  A measure of state anxiety

SECONDARY OUTCOMES:
Chelsea Critical Care Physical Assessment Tool (CPAx) | Assessed at day one
  Measure of physical function
Patient Rehabilitation Satisfaction Questionnaire | 3 weeks post intensive care discharge
  a measure of patient satisfaction with rehabilitation experience

CONTACTS AND LOCATIONS:
Overall Officials: Martina Fitzpatrick, Principal Investigator — Physiotherapy Manager (Temporary), St. Vincent's University Hospital, Elm Park, Dublin 4, Ireland
Locations (1):
- St. Vincent's University Hospital, Dublin, Ireland

REFERENCES:
- [Background] Bench SD, Day TL, Griffiths P. Developing user centred critical care discharge information to support early critical illness rehabilitation using the Medical Research Council's complex interventions framework. Intensive Crit Care Nurs. 2012 Apr;28(2):123-31. doi: 10.1016/j.iccn.2012.02.002. Epub 2012 Mar 3. PMID 22386848